CLINICAL TRIAL: NCT05821231
Title: Phase I Study Evaluating the Safety and Efficacy of MEDI5752 in Combination With Stereotactic Radiotherapy in Patients With Metastatic Sarcoma
Brief Title: Study Evaluating the Safety and Efficacy of MEDI5752 in Combination With Stereotactic Radiotherapy in Patients With Metastatic Sarcoma
Acronym: MEDISARC-SBRT
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: National Cancer Institute, France (Other Government); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21SARC04
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft Tissue Sarcoma; Lung metastasis; Bispecific antibody anti PD-1/CTLA-4; Stereotactic body hypo-fractionated radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with metastatic soft tissue sarcoma with lung metastases (Experimental)
  Interventions: Combination Product: SBRT + MEDI5752

INTERVENTIONS:
Combination Product: SBRT + MEDI5752 — SBRT (5 fractions of 10 Gy every two or three days) will be delivered to one lung metastasis (12 days maximum) in combination with MEDI5752* administered intravenously.
  The first dose of MEDI5752 will be administered on the day of the last SBRT fraction, then every 3 weeks for up to a maximum of 12 months.
  * Dosing 500 mg or 750 mg, according to the recommended dose determined during the dose exploration phase

SUMMARY:
This is a phase I, multicenter, open-label study starting with a dose exploration phase and followed by an expansion phase to evaluate the safety profile and the preliminary activity of the bispecific antibody anti PD-1/CTLA-4 MEDI5752 in combination with SBRT delivered on one lung metastatic lesion, in patients with metastatic soft tissue sarcoma.

Dose exploration phase:

The primary objective of this dose exploration phase I trial is to determine the Maximum Tolerated Dose and the toxicity profile of MEDI5752 when administrated with stereotactic radiotherapy in patients with metastatic sarcoma with lung metastases.

Expansion phase:

The primary objective of the expansion phase is to investigate preliminary activity of MEDI5752 when administrated with stereotactic radiotherapy in patients with metastatic sarcoma with lung metastases.

A maximum of 20 evaluable patients will be included in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed soft tissue sarcoma of following subtype: undifferentiated pleomorphic sarcoma, myxofibrosarcoma, leiomyosarcoma, pleomorphic rhabdomyosarcoma, or pleomorphic liposarcoma
2. Patients with metastatic disease, including (but not restricted to) lung metastasis (in case of lung metastasis only, patients must have more than 5 metastases measurable by RECIST 1.1)
3. Patient with at least two metastases measurable by RECIST 1.1, including at least one lung metastasis amenable for SBRT, defined as following:

   * Tumor size between 1cm and 3 cm, AND
   * Peripheral tumor located further than 2 cm of the proximal bronchial tree (carina, right and left main bronchi, and bronchial tree to the second bifurcation)
4. Metastatic disease pretreated by at least one anthracycline based chemotherapy, but no more than 3 lines of standard therapy
5. Age ≥ 18 years at time of study entry
6. ECOG performance status of 0 or 1
7. Body Weight > 35 kg
8. Life expectancy of at least 3 months
9. Previous treatment ended at least 4 weeks prior to first dose
10. Adequate Hematology laboratory data within 28 days prior to start of treatment: Absolute neutrophils ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hemoglobin ≥ 9 g/dL
11. Adequate Biochemistry laboratory data within 28 days prior to start of treatment: Total bilirubin ≤ 1.5 x ULN (except patient with confirmed Gilbert's syndrome or liver metastasis: Total bilirubin ≤ 3 X ULN), Transaminases ≤ 3 x ULN, Alkalin phosphatases ≤ 5 x ULN, Creatinine clearance ≥ 45 mL/min (Cockcroft)
12. Adequate cardiac function defined as follow: LVEF (as assessed by echocardiography or multiple-gated acquisition scan) ≥ 50% / Troponin I or T ≤ ULN (per institutional guidelines and/or not clinically significant per investigator judgement) / QTcF ≤ 480msec
13. Women should be post-menopaused or willing to accept the use of at least one highly effective method of birth control from screening to 90 days after the last dose of MEDI5752. All non-menopaused women should have a negative pregnancy test within 72 hours prior to study dosing. Men should accept to use an effective contraception from screening to 90 days after the last dose of MEDI5752
14. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
15. Signed written informed consent before any study procedure
16. Patient affiliated to a Social Health Insurance in France

Exclusion Criteria:

1. Patients with no lung metastases amenable for SBRT
2. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to use effective birth control from screening to 90 days after the last dose of MEDI5752
3. Any malignancy other than the disease under study in the past 2 years excepting curatively treated skin cancers such as Basal Cell Carcinoma or Squamous Cell Carcinoma.
4. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed.
5. Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.
6. Severe, active co-morbidity, defined as follows:

   * Unstable angina, uncontrolled cardiac arrhythmia, uncontrolled hypertension, symptomatic congestive heart failure
   * Transmural myocardial infarction within the last 6 months prior to registration
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * Uncontrolled Chronic Obstructive Pulmonary Disease or other respiratory illness requiring hospitalization or precluding study therapy within 30 days prior to registration
   * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
   * History of radiation pneumonitis in the radiation field (fibrosis) is permitted
   * Severe hepatic disease, defined as a diagnosis of Child-Pugh Class B or C hepatic disease
   * Known HIV positive status (positive for HIV-1 or HIV-2 antibodies)
   * End-stage renal disease (i.e., on dialysis or dialysis has been recommended)
   * Active or uncontrolled hepatitis B (HBV) or hepatitis C (HCV). Participants are eligible if they:

     1. Have controlled hepatitis C viral load defined as undetectable hepatitis C RNA by PCR either spontaneously or response to a successful prior course of anti-hepatitis C therapy
     2. Have received HBV vaccination with only anti-HBS positivity and no clinical signs of hepatitis
     3. Are HBsAg- and anti-HBc+ (ie, those who have cleared HBV after infection) and meet conditions i-iii below:
     4. Are HBsAg+ with chronic HBV infection (lasting 6 months or longer) and meet conditions i-iii below:

     i. HBV DNA viral load <100 IU/mL ii. Have normal transaminases values, or, if liver metastases are present, abnormal transaminases, with a result of AST/ALT <3xULN, which are not attributable to HBV infection iii. Start or maintain antiviral treatment if clinically indicated as per the investigator
   * Active hepatitis A
   * Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination, and radiographic findings and TB testing in line with local practice)
7. Active or prior documented autoimmune or inflammatory disorders including inflammatory bowel disease (eg, colitis or Crohn's disease), diverticulitis (with the exception of diverticulosis), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, pneumonitis (past medical history of ILD, drug-induced ILD, or radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD), etc. The following are exceptions to this criterion:

   1. Subjects with vitiligo or alopecia
   2. Subjects with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Subjects with celiac disease controlled by diet alone.
8. History of organ transplant.
9. History of a reaction to any human gamma globulin therapy.
10. Known allergy or hypersensitivity to investigational product, or any excipients of the investigational product
11. Patients with leptomeningeal carcinomatosis
12. Patients with intra cranial metastasis may be eligible if all known lesions have been treated (with stereotactic radiotherapy or surgery or both AND there has been no evidence of disease progression in the CNS for ≥ 4 weeks after treatment and within 28 days prior the first dose of study drug administration
13. Previously Irradiation by SBRT should respect following maximal doses to at-risk structures:

    * Spinal cord irradiated to > 40 Gy
    * Brachial plexus irradiated to > 50 Gy
    * Lung previously with prior V20Gy > 30%
14. Any approved anticancer therapy, including chemotherapy, hormonal therapy or radiotherapy, within 4 weeks prior to initiation of study treatment and while on study treatment; however, the following are allowed: Hormone-replacement therapy or oral contraceptives. Palliative radiotherapy for bone metastases > 2 weeks prior to Cycle 1, Day 1.
15. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI CTCAE v5.0 Grade ≤ 1 or baseline
16. Major surgery within 4 weeks prior to the first dose of investigational product or still recovering from prior surgery. Note: Local surgery of isolated lesions for palliative intent is acceptable
17. Administration of a live, attenuated vaccine within 4 weeks prior to Cycle 1, Day 1. NOTE: Subjects, if enrolled, should not receive live vaccine while receiving investigational product and up to 30 days after the last dose of investigational product
18. Current or prior use of treatment with systemic corticosteroids or other systemic immunosuppressive or immunomodulating medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor [TNF] agents) within 14days prior to the first dose of investigational product. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroids injections (eg. Intraarticular injection)
    2. Steroids as premedication for hypersensitivity reactions (eg CT scan premedication; single palliative dose for pain control etc.)
19. Patient already enrolled in another therapeutic trial involving an investigational substance, and when such a substance has been taken during the previous 4 weeks. The current enrollment in an observational (non interventional) clinical study or the follow-up period of an interventional study is permitted.
20. Prior treatment with PDL-1, PD-1 or CTLA4 blocking agents
21. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Dose exploration Phase: The incidence of the Dose-limiting toxicity (DLT) | 6 weeks after the last dose of radiotherapy for each patient
  For each patient, DLT incidence will be evaluated during the first cycle.
Expansion phase: the rate of patients alive and without progression at 3 months. | 3 months post treatment for each patient

SECONDARY OUTCOMES:
Dose exploration and Expansion Phases: The incidence of Treatment-Emergent Adverse Events will be evaluated using the NCI-CTCAE Version 5.0. | 15 months for each patient
Dose exploration and Expansion Phases: Objective Response Rate (ORR) defined as the rate of patients with an objective response (i.e. CR or PR according to RECIST v1.1 criteria). | 15 months for each patient
Dose exploration and Expansion Phases: Progression-Free Survival (PFS) defined (per RECIST v1.1 criteria) as the time from treatment initiation until progression or death from any cause, whichever occurs first. | 15 months for each patient
Dose exploration and Expansion Phases: Time to progression of irradiated lesions defined as the time from treatment initiation until progression of irradiated lesions or death from any cause. | 15 months for each patient
Dose exploration and Expansion Phases: Time to progression outside the irradiation field defined as the time from treatment initiation until progression outside the irradiation field or death from any cause. | 15 months for each patient
Dose exploration and Expansion Phases: Overall Survival (OS) defined as the time from treatment initiation to death from any cause. | 15 months for each patient

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Regional Du Cancer de Montpellier, Montpellier
  - IUCT-O, Toulouse